CLINICAL TRIAL: NCT05154916
Title: The Effect of Virtual Reality-Based Relaxation Program on Pain Severity, Anxiety Level and Patient Satisfaction in Patients to be Performed Bronchoscopy
Brief Title: The Effect of Virtual Reality Based Relaxation Program on Patients to be Performed Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, gülcan bahcecioğlu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E-97132852-050.01.04-87889
Record Dates: First submitted 2021-11-18; First posted 2021-12-13 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Bronchoscopy; Virtual Reality; Glasses; Relaxation Program

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: (Experimental): Bronchoscopy of Virtual Reality Based Relaxation Program Will Be Applied
  Interventions: Other: Virtual Reality Based Relaxation Program
- No Intervention (No Intervention): Bronchoscopy of Virtual Reality Based Relaxation Program Will Not Be Applied

INTERVENTIONS:
Other: Virtual Reality Based Relaxation Program — Virtual Reality Based Relaxation Program
  Arms: Experimental:

SUMMARY:
With the virtual reality application in patients with bronchoscopy, it is aimed to reduce the fear, stress and tension arising from the possibility of the development of pain and complications in the patients. The research will be carried out in the form of pretest-posttest application with 30 experimental and 30 control groups. The researcher aims to minimize the fear and stress in the patient by applying the virtual reality application to the patient in the experimental group 10 minutes before the procedure and 5-10 minutes during the procedure. The researcher will download the licensed program called 'a walk on the beach' to the virtual reality glasses and the patient will watch this program with glasses. The patient in the experimental group will have to fill in the Visual Analogue Scale, Anxiety Evaluation Form, Anxiety Symptoms Follow-up Form, and Patient Information Form before the procedure. 10-15 minutes after the procedure, the patient will be asked to fill the Visual Analogue Scale, Anxiety Evaluation Form, Anxiety Symptoms Follow-up Form and the Virtual Reality Glasses Application Satisfaction Form. No procedure will be applied to the patients in the control group and they will be asked to fill in the Patient Information Form, Visual Analogue Scale Form, Anxiety Evaluation Scale Form, and Anxiety Symptoms Follow-up Form before the procedure. After the procedure, he will be asked to fill in the other forms again, except the Patient Information Form. Patients over the age of 18, who have no communication problems, no psychiatric problems, who volunteered to participate in the study, and who had local application in bronchoscopy will be included in the study. Patients with psychiatric problems and communication problems will not be included in the study. Before the procedure, the patient will be informed that his/her identity information will be kept confidential and that he/she can withdraw from the research at any time, and all his/her rights will be informed.

DETAILED DESCRIPTION:
This study includes the examination of the effect of applying virtual reality interventions, which are used for the treatment of anxiety problems, to patients who will undergo bronchoscopy. For this purpose, first of all, a relaxation intervention will be designed in a virtual reality environment. The virtual reality environment will be organized on the basis of relaxation exercise. In this direction, first of all, an image will be created by taking 3D modeling service and the text of the relaxation exercise prepared in the presence of a professional sound artist will be transferred to the image with sound. Afterwards, the relaxation exercise created will be applied to the patients before and during the bronchoscopy application. The aim of this study; It is aimed to examine the Effect of Virtual Reality Based Relaxation Program on Pain Severity, Anxiety Level and Patient Satisfaction in Patients to be Performed Bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* be18 years and over
* Ability to communicate adequately
* Absence of psychiatric problems
* Those who are determined by the physician that they do not have a physical disability in exercising
* Volunteering to participate in the research
* Individuals who have the ability to use technological tools
* Patients who underwent local application in bronchoscopy

Exclusion Criteria:

* Those who have communication problems
* Those with psychiatric problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale Evaluation | 60 minutes
  Visual Analog Scale is used to convert some values that cannot be measured numerically into digital. Two end definitions of the parameter to be evaluated are written at the two ends of a 100 mm line and the patient is asked to indicate where on this line their situation is appropriate by drawing a line or by placing a dot or pointing.0 points means no pain, 100 points means a lot of pain
Virtual Reality Glasses Application Satisfaction Form | 60 minutes
  In this form, there are questions prepared in line with the relevant literature (Dutucu, 2019) in order to determine the satisfaction with the video watched with virtual reality glasses.The higher the score, the higher the satisfaction
Anxiety Assessment Scale | 60 minutes
  Patients will be asked to show their anxiety levels before and after the procedure on a 10 cm long horizontal line. Line has 0 at the beginning and 10 at the end. 10 means very extreme anxiety and 0 means no anxiety.
Physiological Symptoms of Anxiety Follow-up Form | 60 minutes
  This form was created by the researcher to record blood pressure, heart rate, respiratory rate and peripheral oxygen saturation value.These values will be checked again in 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Gülcan B Turan, Study Chair — Firat University
Locations (1):
- Fırat university, Elâzığ, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No